CLINICAL TRIAL: NCT06961578
Title: Surgical Versus Conservative Treatment of Odontoid Fractures in the Elderly: A Randomised Controlled Clinical Study (SCORE)
Brief Title: SCORE Study: Comparing Surgery and Rigid Collar Treatment for Odontoid Fractures in Adults Over 70
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: St. Josefs-Hospital Wiesbaden GmbH (Other); Medical University of Cologne (Other); BG Trauma Center Tuebingen (Other); RWTH Aachen University (Other); University Hospital Heidelberg (Other); University Hospital, Essen (Other); BG Klinikum Bergmannstrost, Halle, Germany (Unknown); Helios Klinikum Berlin-Buch (Other); German Federal Ministry of Education and Research (Other Government); Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-630-S-NP; 01KG2405 (Other Grant/Funding Number: German Federal Ministry of Education and Research, BMBF)
Record Dates: First submitted 2025-04-20; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Odontoid Fracture; Elderly
Keywords: Odontoid fracture; C2 fracture; atlantoaxial instability; atlantoaxial fusion; Barthel Index; functional outcome
MeSH Terms: conditions — Atlanto-Axial Fusion | interventions — Spinal Fusion; Gene Fusion

STUDY DESIGN:
Intervention Model Description: Two-arm, prospective, multi-center, open-label, randomized, controlled non-inferiority clinical study in a parallel group design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservative Group (Experimental): conservative group subjected to external collar bracing
  Interventions: Other: External immobilization with rigid cervical collar
- Surgical Group (Experimental): surgical group undergoing C1-2 instrumentation
  Interventions: Procedure: C1-2 instrumentation

INTERVENTIONS:
Procedure: C1-2 instrumentation — Surgical fracture stabilization with a posterior screw-rod system from C1-2 from a posterior approach.
  The routine surgery commonly lasts approximately 100 minutes and requires a hospital stay of about 6 days. An additional external bracing in the postoperative setting is not required.
  Other Names: Spondylodesis; fusion
  Arms: Surgical Group
Other: External immobilization with rigid cervical collar — External immobilization with a rigid cervical collar for 12 weeks. Compliance is monitored through patient diaries, recognizing the real-world challenges of consistent brace use. Lack of adherence is considered to reflect routine clinical practice. A typical drawback of the conservative intervention in daily practice is the absolute reliance on patient compliance to wear the collar continuously for at least 12 weeks, which poses a significant challenge to this treatment strategy.
  Arms: Conservative Group

SUMMARY:
The goal of this clinical trial is to compare two treatment options-surgery or rigid collar bracing-for unstable neck fractures (odontoid fractures) in adults aged 70 years and older. These fractures are common in older adults and can significantly impact mobility, independence, and quality of life. There is currently no clear evidence to determine which treatment is better for this population. The main questions it aims to answer are:

* Does surgery or conservative collar treatment lead to better improvement in daily living, measured by the Barthel Index, after 12 weeks?
* What are the differences in pain, disability, and quality of life between the two treatments?

The study team will compare patients who receive surgical stabilization with those who are treated with a rigid cervical collar to see which approach supports better functional outcomes and healing.

Participants will:

* be randomly assigned to either surgery (posterior C1-C2 screw-rod fixation) or conservative collar treatment
* attend study visits at 12 weeks and 6 months
* complete questionnaires on daily functioning, pain, and quality of life
* undergo CT scans and other medical assessments
* record collar use (for conservative group) in a diary
* be monitored for any complications or changes in treatment (including crossover to surgery if needed)

The study aims to include 322 participants to provide evidence on which treatment helps older adults recover better from odontoid fractures with fewer complications and improved quality of life.

DETAILED DESCRIPTION:
The SCORE study is a multicenter, randomized, controlled, open-label, parallel-group non-inferiority trial designed to provide evidence on whether conservative treatment is non-inferior to surgical stabilization regarding recovery of daily functioning.

Study Objectives A) Primary Objective: To compare the effectiveness of surgical versus conservative treatment for unstable OFs in patients aged 70 or older in terms of recovery in activities of daily living, measured by the change in Barthel Index (BI) from baseline to 12 weeks.

B) Secondary Objectives: To compare the effects of treatment on:

* Quality of life (EQ-5D)
* Neck pain (Visual Analog Scale)
* Neck-specific disability (Neck Disability Index)
* Radiographic fracture healing
* Treatment compliance
* Rate of crossover from conservative to surgical treatment
* Incidence of adverse and serious adverse events

This is a prospective, two-arm, multicenter, randomized controlled non-inferiority trial with parallel-group design. Patients will be randomized 1:1 to receive either surgical stabilization (posterior C1-C2 screw-rod fixation) or conservative treatment with a rigid cervical collar. Randomization will be stratified by center using permuted blocks via the secure online platform randomizer.at. Participants are followed up at 12 weeks and 6 months post-injury. An additional visit ~2 weeks after surgery is conducted for those undergoing surgical treatment. Patients in the conservative arm may cross over to surgery up to week 12, based on clinical indication or patient preference.

Intervention Descriptions A) Surgical Group: Posterior stabilization using a screw-rod system without additional external bracing. The surgery lasts ~100 minutes and requires ~6 days of hospital stay. This approach is tailored for geriatric patients and excludes anterior fixation due to biomechanical concerns in the elderly.

B) Conservative Group: External immobilization using a rigid cervical collar for 12 weeks. Compliance is monitored via patient diaries, acknowledging real-world challenges in consistent brace use. Lack of adherence is considered reflective of routine clinical practice.

Statistical Analyses The primary analysis will assess non-inferiority of conservative treatment versus surgery using a mixed model for repeated measures (MMRM) of the BI at 12 weeks. Covariates include treatment, time, interaction terms, baseline BI, age, and CCI; study center is treated as a random effect (excluded if convergence fails). Non-inferiority is defined by a margin of 5 BI points, which is more conservative than the minimal clinically important difference (MCID) of 9.8 and closer to the smallest detectable change (SDC) of 3.0, based on prior studies. The study has 90% power to detect non-inferiority (one-sided α = 0.025). A total of 137 patients per arm (274 total) are needed, inflated to 322 to account for 15% attrition.

Secondary analyses will use similar mixed models for continuous variables and generalized estimating equations for binary outcomes. Sensitivity analyses include "as-treated" models accounting for crossover. No adjustment for multiple comparisons will be made.

Randomization Procedure Randomization is conducted after informed consent via randomizer.at. Lists are stratified by center and use permuted blocks. Access is password-protected and managed by study personnel.

An independent Data and Safety Monitoring Board (DSMB) will oversee the study. All adverse events and serious adverse events are recorded at each visit and coded per MedDRA prior to analysis.

ELIGIBILITY:
Inclusion Criteria:

* At least 70 years old
* Acute unstable OFs (types II, III as classified by Anderson and d'Alonzo, and atypical)
* Less than two weeks post injury
* Written informed consent

Exclusion Criteria:

* Previous treatment for odontoid fracture
* Concomitant fractures of the subaxial cervical spine necessitating surgery
* Significant comorbidity resulting in inoperability of the patient: i.e. ASA score > 4
* Neurological compromise due to displaced fracture

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 322 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-12-12 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Barthel Index | Baseline to 12 weeks
  Change in Barthel Index (BI) between baseline and 12 weeks thereafter

SECONDARY OUTCOMES:
Change in quality of life assessed by the EuroQol 5 Dimensions (EQ-5D) | Baseline to 12 weeks and to 6 months.
  Change in quality of life assessed by the EQ-5D between baseline, 12 weeks and 6 months. Minimum score 0, Maximum score 100, higher scores denote higher perceived quality of life.
Duration of surgery | Baseline value (time of surgery)
  Duration of surgery for the surgery/intervention group.
Duration of time per day the cervical collar is worn (patient/proxy protocol) | Baseline to 12 weeks
  Duration of time per day the cervical collar is worn (patient/proxy protocol)
Neck-Disability-Index (NDI) | Baseline, 12 weeks and 6 months after surgery/intervention
  Patient-completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation.
Charlson Comorbidity Index (CCI) | Baseline value
  Charlson Comorbidity Index predicts the ten-year mortality for a patient who may have a range of comorbid conditions.
Union rate of fracture | 12 weeks after surgery/intervention
  Union rate of fracture assessed by CT scan after 12 weeks
Readmission to hospital | Baseline to 12 weeks to 6 months
  Readmission to hospital from baseline to 12 weeks to 6 months.
Cross-over rate | Baseline to 12 weeks
  Cross-over rate from conservative to surgical arm
Change in Visual Analogue Scale Pain (VAS) | baseline, immediately after surgery/intervention, 12 weeks after surgery/intervention and 6 months after surgery/intervention
  Change in VAS between baseline, postoperative/at discharge (5 - 14 days post surgery), 12 weeks and 6 months after surgery/intervention

CONTACTS AND LOCATIONS:
Locations (16):
- Germany (16):
  - LMU University Hospital, Munich, Bavaria
  - Center for Spinal Surgery and Neurotraumatology, Berufsgenossenschaftliche Unfallklinik, Frankfurt am Main, Hesse
  - Department of Neurosurgery, RWTH Aachen University, Aachen
  - Charité University Hospital Berlin, Berlin
  - Department of Neurosurgery and Spine Center, HELIOS Hospital Berlin Buch, Berlin
  - Department of Orthopaedic and Traumatology, University of Cologne, Cologne
  - Department of Orthopedics, Medical University at Dresden, Dresden
  - Department of Neurosurgery and Spine Surgery, University Hospital Essen, Essen
  - Department of Neurosurgery, University Medical Center Göttingen, Göttingen
  - Department of Trauma and Reconstructive Surgery, BG Klinikum Bergmannstrost Halle, Halle
  - Department of Neurosurgery, University Hospital Heidelberg, Heidelberg
  - Department of Neurosurgery, University Hospital of Lausitz, Lausitz
  - Department of Orthopaedics, Trauma Surgery and Plastic Surgery, University of Leipzig, Leipzig
  - Spine Surgery, Orthopedic Hospital Markgröningen GmbH, Markgröningen
  - BG Trauma Centre, Eberhard Karls University of Tuebingen, Tübingen
  - Spine Center, St. Josefs-Hospital Wiesbaden, Wiesbaden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wagner A, Albrecht C, Dittmer S, Egert-Schwender S, Kehl V, Stichling R, Klatt G, Ettinger B, Hecht N, Vajkoczy P, Wengert A, Kandziora F, von der Hoh NH, Heyde CE, Hartung P, Richter M, Lenz M, Eysel P, Badke A, Blume C, Clusmann H, Walter J, Krieg S, Evangelou P, Shiban E, Dreimann M, Gembruch O, Sure U, Bettag C, Rohde V, Disch A, Bekele B, Ryang YM, Kramer A, Ringel F, Wach J, Guresir E, Meyer B, Wostrack M. Surgical versus conservative treatment of odontoid fractures in the elderly: A randomized controlled clinical study (SCORE). PLoS One. 2025 Dec 23;20(12):e0337999. doi: 10.1371/journal.pone.0337999. eCollection 2025. PMID 41433244